CLINICAL TRIAL: NCT07076095
Title: A Phase II/III Study to Compare IBB0979 in Combination With Topotecan Versus Topotecan in Subjects With Relapsed Small Cell Lung Cancer
Brief Title: A Phase II/III Study of IBB0979 in Combination With Topotecan Versus Topotecan in Relapsed Small Cell Lung Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: SUNHO（China）BioPharmaceutical CO., Ltd. (Industry)
Collaborators: The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBB0979-201
Record Dates: First submitted 2025-07-17; First posted 2025-07-21 (Actual); Last update posted 2025-07-21 (Actual); Status verified 2025-07

CONDITIONS: Small Cell Lung Cancer
MeSH Terms: conditions — Small Cell Lung Carcinoma | interventions — Topotecan; Injections

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Part 1(Phase IIa) (Experimental): To evaluate the safety and efficacy of IBB0979 in patients with SCLC. Cohort 1: IBB0979 iv Q3W; Cohort 2: IBB0979 iv Q2W.
  Interventions: Drug: IBB0979
- Part 2(Phase IIb) (Experimental): To evaluate the safety and efficacy of IBB0979 in combination with topotecan in patients with SCLC.
  Interventions: Drug: IBB0979; Drug: topotecan hydrochloride for injection

INTERVENTIONS:
Drug: IBB0979 — bifunctional antibody-cytokine fusion protein that targets B7-H3 and IL-10 receptor
Drug: topotecan hydrochloride for injection — Topotecan hydrochloride will be administered intravenously per prescribing information.
  Arms: Part 2(Phase IIb)

SUMMARY:
This study was designed to compare the efficacy and safety of IBB0979 in combination with topotecan versus topotecan in subjects with relapsed small cell lung cancer (SCLC).

ELIGIBILITY:
Inclusion Criteria:

1. Aged ≥18 and ≤75 years, male or female.
2. Histologically confirmed SCLC.
3. Relapsed small cell lung cancer (limited-stage, extensive-stage) that has failed or progressed after first-line or second-line systemic therapy.
4. At least one measurable lesion according to RECIST version 1.1.
5. ECOG PS 0 or 1.
6. Life expectancy ≥ 3 months.
7. Adequate organ function.
8. Men or women should be using adequate contraceptive measures throughout the study. Females subjects must not be pregnant at screening or have evidence of non-childbearing potential.
9. Signed and dated Informed Consent Form.

Exclusion Criteria:

1. Combined SCLC, any previous diagnosis of transformed SCLC or SCLC that has transformed to NSCLC.
2. Known hypersensitivity (≥ Grade 3) to recombinant proteins or any excipient contained in the drug or vehicle formulation for IBB0979.
3. History of anti-tumor therapy (chemotherapy, radiotherapy, biological therapy, endocrine therapy, targeted therapy within 4 weeks) prior to the initiation of investigational product administration.
4. History of any un-marketed investigational product or therapy within 4 weeks prior to the initiation of investigational product administration.
5. History of major organ surgery (with exception of aspiration biopsy) or significant trauma within 4 weeks prior to the initiation of investigational product administration, or selective operation is required during the trial.
6. History of systemic corticosteroid therapy with exceptions defined in the protocol.
7. Treatment with immunomodulatory agents, including but not limited to thymosin, interleukin-2 and interferon within 14 days prior to the initiation of investigational product administration.
8. Vaccination with any live virus vaccine within 4 weeks prior to the initiation of investigational product administration.
9. History of prior allogeneic stem-cell or solid organ transplantation.
10. Unresolved toxicity from prior anti-tumor therapy, defined as not having resolved to Common Terminology Criteria for Adverse Events (CTCAE) version 5.0 grade 1 with exceptions defined in the protocol.
11. Untreated brain metastases with exceptions defined in the protocol.
12. Evidence of active infection requiring intravenous anti-infective therapy.
13. Have a history of immune deficiency, including a positive test for human immunodeficiency virus (HIV) antibodies.
14. Active hepatitis B, active hepatitis C.
15. Currently has interstitial lung disease (with exception of radiation pulmonary fibrosis that requires no hormone therapy).
16. History of severe cardiovascular and cerebrovascular diseases.
17. Active or suspected autoimmune diseases (such as systemic lupus erythematosus, rheumatoid arthritis, vasculitis, etc.) with exceptions defined in the protocol.
18. History of ≥ grade 3 immune-related adverse events (irAE) or Grade 2 immune-associated myocarditis accompanied with immunotherapy with exceptions defined in the protocol.
19. History of other malignancy with exceptions defined in the protocol.
20. Pleural effusion/peritoneal effusion/Pericardial effusion requiring clinical intervention.
21. Known alcohol or drug dependence.
22. History of mental disorder or poor adherence.
23. The female patient who is pregnant or breastfeeding.
24. History of other severe systemic disease, or any issue that in the opinion of the investigator, would contraindicate the patient's participation in the study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2028-08-01 (Estimated); Study Completion 2031-08-01 (Estimated)

PRIMARY OUTCOMES:
Frequency of adverse events (AEs) and SAEs (Phase II) | Approximately within 36 months
  To investigate the safety characteristics.

SECONDARY OUTCOMES:
Pharmacokinetic (PK) Cmax (Phase II) | Approximately within 36 months
  PK parameters (Cmax) following single dose.
Pharmacokinetic (PK) Cmin (Phase II) | Approximately within 36 months
  PK parameters (Cmin) following single dose.
Pharmacokinetic (PK) Tmax (Phase II) | Approximately within 36 months
  PK parameters (Tmax) following single dose.
Pharmacokinetic (PK) AUC 0-t (Phase II) | Approximately within 36 months
  PK parameters (AUC 0-t) following single dose.
Pharmacokinetic (PK) AUC 0-∞ (Phase II) | Approximately within 36 months
  PK parameters (AUC 0-∞) following single dose.
Pharmacokinetic (PK) CL (Phase II) | Approximately within 36 months
  PK parameters (CL) following single dose.
Pharmacokinetic (PK) Vd (Phase II) | Approximately within 36 months
  PK parameters (Vd) following single dose.
Pharmacokinetic (PK) t1/2 (Phase II) | Approximately within 36 months
  PK parameters (t1/2) following single dose.
Pharmacokinetic (PK) λz (Phase II) | Approximately within 36 months
  PK parameters (λz) following single dose.
Pharmacokinetic (PK) Css,max (Phase II) | Approximately within 36 months
  PK parameters (Css,max) following multiple dose.
Pharmacokinetic (PK) Css,min (Phase II) | Approximately within 36 months
  PK parameters (Css,min) following multiple dose.
Pharmacokinetic (PK) Css,av (Phase II) | Approximately within 36 months
  PK parameters (Css,av) following multiple dose.
Pharmacokinetic (PK) AUCss (Phase II) | Approximately within 36 months
  PK parameters (AUCss) following multiple dose.
Pharmacokinetic (PK) CLss (Phase II) | Approximately within 36 months
  PK parameters (CLss) following multiple dose.
Pharmacokinetic (PK) Vss (Phase II) | Approximately within 36 months
  PK parameters (Vss) following multiple dose.
Pharmacokinetic (PK) R (Phase II) | Approximately within 36 months
  PK parameters (R) following multiple dose.
Pharmacokinetic (PK) DF (Phase II) | Approximately within 36 months
  PK parameters (DF) following multiple dose.
Incidence of Anti-Drug Antibodies (ADA)(Phase II) | Approximately within 36 months
Overall survival (OS) (Phase II) | Baseline through up to 2 years or until disease progression
  OS as assessed using RECIST 1.1.
Objective response rate (ORR)(Phase II) | Baseline through up to 1 years or until disease progression
  Tumor response based on RECIST 1.1.
Progression free survival (PFS) (Phase II) | Baseline through up to 2 years or until disease progression
  PFS as assessed using RECIST 1.1.
Disease control rate (DCR) (Phase II) | Baseline through up to 2 years or until disease progression
  DCR as assessed using RECIST 1.1.

CONTACTS AND LOCATIONS:
Overall Officials: ming qi wang, Principal Investigator — The Affiliated Cancer Hospital of Zhengzhou University & Henan Cancer Hospital